CLINICAL TRIAL: NCT01210027
Title: A Pilot Study of Radiation Toxicity in the Liver Using MRI-Based Perfusion
Brief Title: A Study of Radiation Toxicity in the Liver Using MRI-Based Perfusion
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2006.067; HUM 5910 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2010-09-02; First posted 2010-09-28 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Researchers at the the University of Michigan are conducting a research project to assess how a course of radiation therapy changes the way blood flows through the liver. To be able to do this, the researchers will be using MRI (magnetic resonance imaging) scans completed before, during, and after radiation therapy. MRI's will be done on 4 or 5 occasions. On each occasion, you will be injected with a fluid called gadolinium (a contrast agent) before getting an MRI. This contrast agent makes it easier for the Researchers to see your organs in the scans, and causes any abnormal areas to become very bright on the MRI. This agent will be injected into a vein in your arm or leg. Each MRI scan will last approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥18 years of age.
* The patient's planned cancer management is radiation to the liver with or without chemotherapy.
* Patients must have a performance status of 0-2 and a life expectancy of at least 3 months.
* Patients should have no contraindications to having a contrast enhanced MRI scan.

Exclusion Criteria:

* Women who are pregnant or breastfeeding are excluded.
* Prisoners are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have one of the following: primary hepatocellular cancer, hepatobiliary cancer, or metastatic disease to the liver.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Measure of Liver Function Before, During and After Radiation | 2-3 months for treatment; indefinite for follow-up
  The primary objective of this research is to assess how a course of radiation therapy changes the way blood flows through the liver. Researchers want to use the information collected from this research for future research, to see if this change in blood flow indicates that an individual patient is at higher risk for complications from the radiation therapy, specifically Radiation-Induced Liver Disease (RILD). To be able to do this, the researchers will be using MRI (magnetic resonance imaging) scans completed before, during, and after radiation therapy.

SECONDARY OUTCOMES:
Measure of Liver Perfusion | Follow-up - Approximately 7 Years
  Develop a model to predict post-treatment liver perfusion based on pre-treatment perfusion, intratreatment perfusion, and radiation dose.
Association Between Liver Perfusion and Changes in Tumor and Clinical Outcomes | Follow-up - Approximately 7 years
  Explore the association between liver perfusion changes in tumor and clinical outcomes, including the size of tumor; local tumor progression; distant metastases; overall survival; and toxicity (radiation-induced liver disease).

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lawrence, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States